CLINICAL TRIAL: NCT00659841
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase 3 Clinical Trial to Assess the Safety and Efficacy of Ciclesonide, Applied as a Nasal Spray (200µg Once Daily) in the Treatment of Seasonal Allergic Rhinitis (SAR) in Patients 12 Years and Older
Brief Title: To Assess the Safety and Efficacy of Ciclesonide, Applied as a Nasal Spray in the Treatment of Seasonal Allergic Rhinitis (BY9010/M1-401)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY9010/M1-401
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Seasonal; Hay Fever
Keywords: Seasonal Allergic Rhinitis; Ciclesonide; Hay Fever; SAR
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): Ciclesonide 200µg
  Interventions: Drug: Ciclesonide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide — 200µg Ciclesonide versus placebo
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of ciclesonide applied as a nasal spray once daily in patients with SAR. The secondary objectives are to evaluate Quality-of-Life and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 12 years and older.
2. General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the trial.
3. A history of SAR to relevant seasonal allergen for a minimum of two years immediately preceding the study season. The SAR must have been of sufficient severity to have required treatment (continuous or intermittent) in the past and in the investigator's judgment, - is expected to require treatment throughout the entire study period.
4. A demonstrated sensitivity to Mountain Cedar pollen known to induce SAR through a standard prick test. A positive test is defined as a wheal diameter at least 3 mm larger than the control wheal for the prick test. Documentation of a positive result 12 months prior to screening is acceptable.
5. Female is of child-bearing potential and is currently taking and will continue to use a medically reliable method of contraception for the entire study duration (e.g. oral, injectable, trans-cutaneous or implantable contraceptives or intrauterine devices or double-barrier protection). Women of childbearing potential, or less than 1 year postmenopausal, will require a negative serum pregnancy test at the Screening Visit (B0) as well as at last on-treatment visit (T4).
6. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and compliance with all study requirements (visits, record keeping, etc).

Exclusion Criteria:

1. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the study period.
2. History or physical findings of nasal pathology, including nasal polyps within the last 60 days) or other clinically significant respiratory tract malformations, recent nasal biopsy (within the last 60 days), nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa (within the last 60 days).
3. Participation in any investigational drug trial within the 30 days preceding the Screening Visit.
4. A known hypersensitivity to any corticosteroid or any of the excipients in the formulation.
5. History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, the common cold, acute or chronic sinusitis, flu, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit, or development of a respiratory infection during the Screening Period.
6. History of alcohol or drug abuse within the preceding two years.
7. History of a positive test for HIV, hepatitis B or hepatitis C.
8. Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of b-agonists; intermittent use of b-agonists is acceptable.
9. Plans to travel outside the study area (the known pollen area for the investigative site) for two or more consecutive days OR 5 or more days total during the 5-week study period ( Baseline and Treatment Periods).
10. Use of any prohibited concomitant medications within the prescribed (per protocol) time since last dose period prior to the Screening Visit (B0) and during entire treatment duration.
11. Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit (B0). Low doses of antibiotics taken for prophylaxis are permitted if the therapy was started prior to the Screening Visit AND is expected to continue throughout the trial.
12. Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit AND use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
13. Previous participation in an intranasal ciclesonide study.
14. Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit (B0).
15. Exposure to systemic corticosteroids for any indication, chronic or intermittent (e.g.: contact dermatitis), during the past 2 months, or presence of an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
16. Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone for dermatological conditions during the past 1 month, or presence of an underlying condition that can reasonably be expected to require treatment with such preparations during the course of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2003-12; Primary Completion 2004-12 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Average of AM and PM patient-reported reflective Total Nasal Symptom Score (TNSS) over the first two weeks of treatment | 4 weeks

SECONDARY OUTCOMES:
Instantaneous patient-reported TNSS over the first two weeks of treatment | 4 weeks
Physician Assessment of Overall Nasal Signs and Symptoms Severity (PANS) at Endpoint | 4 weeks
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) at Endpoint | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (4):
- United States (4):
  - Altana/Nycomed, Austin, Texas
  - Altana/Nycomed, Kerrville, Texas
  - Altana/Nycomed, New Braunfels, Texas
  - Altana/Nycomed, San Antonio, Texas

REFERENCES:
- See also: BY9010-M1-401-RDS-2004-12-21.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4529&filename=BY9010-M1-401-RDS-2004-12-21.pdf